CLINICAL TRIAL: NCT03209895
Title: A Double-Blinded, Placebo Controlled, Human Clinical Study to Evaluate the Safety and Efficacy of a Proprietary "Joint Health" Dietary Supplement in Subjects With Joint and Connective Tissue Pain
Brief Title: Study to Evaluate the Safety and Efficacy of a Proprietary "Joint Health" Dietary Supplement in Subjects With Joint and Connective Tissue Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Nutraceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KO1
Record Dates: First submitted 2017-06-29; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia | interventions — Glucosamine; Chondroitin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Joint Health Product (Experimental)
  Interventions: Dietary Supplement: Joint Health Product
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Glucosamine / Chondroitin (Active Comparator)
  Interventions: Dietary Supplement: Glucosamine / Chondroitin

INTERVENTIONS:
Dietary Supplement: Joint Health Product — Krill oil, Astaxanthin, Hyaluronic Acid Formulation, 353 mg per day; Softgel capsule
  Other Names: FlexPro MD
  Arms: Joint Health Product
Dietary Supplement: Placebo — Palm oil Softgel capsule
  Arms: Placebo
Dietary Supplement: Glucosamine / Chondroitin — Glucosamine 1500 mg, Chondroitin 1200 mg per day
  Arms: Glucosamine / Chondroitin

SUMMARY:
This study is designed to evaluate the effectiveness of a proprietary nutritional supplement that contains Krill Oil (KO), astaxanthin (AX) and hyaluronic acid (HA) to reduce pain and discomfort in participants, compared to an inert placebo (palm oil) control and to a positive control (glucosamine-chondroitin). The purpose of the study is to determine if the combination of KO, AX, and HA will benefit participants with joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able and willing to give Informed Consent.
* Subjects must not have taken anti-inflammatory drugs or supplements for 5 days prior to their initial C-RP blood test, and must refrain from taking these products for the duration of the study.
* Subjects will be required to refrain from taking other pain-reducing agents during the course of the study. This will ensure that the effects observed in the study are the effects of the supplement only, and not of other anti-inflammatory agents
* Subjects must have had knee or hip joint or muscle pain on most days of the previous month; should not have "morning stiffness" for more than 30 minutes; and should experience "stiffness" after resting.
* Subjects must have persistent pain in the knee or hip joints or connective tissue with a pain assessment score of at least 5, but not more than 9 using the WOMAC Pain Assessment and Pain Intensity Rating scale.
* Subjects must be available for and willing to attend all evaluation visits.
* Subjects must be willing to take/use the test Krill Oil compositions in place of current pain relief medications.
* Subjects may not be on any steroid-based therapies.
* Subjects must have access to a telephone for calling into the Clinical Center as part of test product compliance.
* Subjects must be willing to use appropriate birth control for duration of trial (if appropriate)
* Subjects must be willing to limit consumption of fatty fish for one week prior to and during the study
* Subjects must be willing to refrain from taking any other nutritional supplements related to immune function or pain reduction during the course of this study.

Exclusion Criteria:

* Subjects must not be taking remission-inducing drugs such as methotrexate.
* Subjects whose joint pain is not in their knees.
* Subjects who are not willing to forego the use of anti-inflammatory and anti-pain medications or supplements for the duration of the study.
* Subjects who know that their joint pain is due to osteoarthritis or rheumatoid arthritis.
* Women who are pregnant, breastfeeding, or planning to become pregnant during the
* course of the trial
* Clinical evidence or known history of severe cardiac, pulmonary, gastrointestinal, renal, hepatic or neurological disorders.
* History of allergy to aspirin or NSAlDs.
* Subjects who have undergone total knee replacement in the contra-lateral knee within 6 months prior to the screening visit.
* Subjects who have received an intra-articular corticosteroid injection in a lower joint during the three (3) months prior to the baseline visit.
* Subjects with isolated lateral compartment disease defined by joint space loss in the lateral compartment only.
* Subjects who have received chondrocyte transplants in any lower extremity joint.
* Subjects with co-morbid conditions that restrict knee function.
* Treatment with corticosteroids before washout period
* Patients with infectious arthritis or gout
* Unstable medical conditions.
* Use of omega fatty acid supplements within two weeks of this study
* Clinically significant abnormal laboratory results at baseline
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy, especially from crustaceans, or sensitivity to study supplement ingredients
* Individuals cognitively impaired and/or who are unable to give Informed Consent
* Any other health or mental condition that in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or that may pose significant risk to the subject
* Subjects taking Inflammatory medications, cardiovascular medications, hypotensive medications, blood thinners
* Presence of auto immune diseases, other diseases of the immune systems,
* gastrointestinal diseases, i.e. Irritable bowel syndrome, or disorders of lipid metabolism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-10-08 (Actual); Primary Completion 2011-06-13 (Actual); Study Completion 2011-06-13 (Actual)

PRIMARY OUTCOMES:
WOMAC Change | Days: 0, 14, 28 and 56
  Change in Clinical Coordinator administered pain assessment and pain intensity evaluation over 56 days as determined by the Western Ontario and McMaster Universities Osteoarthritis Index™© (WOMAC)
VAS Change | Days: 0, 7, 14, 28, 35, 42 and 56
  Change in Self-administered Visual Analogue Pain Assessment and Pain Intensity Rating Scale (VAS) over 56 days

SECONDARY OUTCOMES:
Blood Chemistry CBC Change | Days: 0, 14, 28 and 56
  Change in CBC and differentials over 56 days
Blood Chemistry hs-CRP Change | Days: 0, 14, 28 and 56
  Change in hs-CRP over 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Eshwari Koovor, M.B.B.S., Principal Investigator — PI; Herjit Pannu, MD, Principal Investigator — PI
Locations (1):
- 1621 Bridgeway, Sausalito, California, United States

IPD SHARING:
Plan to Share IPD: No